CLINICAL TRIAL: NCT02299843
Title: A Prospective Randomized Controlled Trial of Radio-frequency Assisted ALPPS（RALPPS）and Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy（ALPPS）in the Treatment of Hepatocellular Carcinoma.
Brief Title: RALPPS Venus ALPPS for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Jun, institute of hepatobiliary surgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014KYNO.51
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: RFA; ALPPS; hepatectomy; morbidity and mortality
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALPPS (Active Comparator): Using ALPPS for the the treatment of hepatocellular carcinoma.
  Interventions: Procedure: ALPPS
- RALPPS (Experimental): Using radiofrequency ablation instead of in-situ split of liver in ALPPS stage I（RALPPS）.Habib 4X was used in RFA.
  Interventions: Procedure: RALPPS

INTERVENTIONS:
Procedure: RALPPS — Using radiofrequency ablation assisted ALPPS（RALPPS）instead of in-situ split of liver to form a coagulation band in stage I.Habib 4X was used in RFA.
  Arms: RALPPS
Procedure: ALPPS — Treat the hepatocellular carcinoma with ALPPS.
  Arms: ALPPS

SUMMARY:
Currently，the "ALPPS" (associating liver partition with portal vein ligation for staged hepatectomy) procedure which enables the rapid growth of the future liver remnant and extends surgical indication to patients with mid-advanced stage hepatocellular carcinoma becomes a research hot spot. However, the procedure has a high morbidity and mortality rate.Using radio-frequency ablation instead of in-situ split of liver to avoid forming a coagulation band in stage I will reduce the incidence of complications（bile leakage, abdominal infection,hemorrhage e.t.) The investigators named this technique as Radio-frequency Assisted Liver Partition with Portal vein ligation for staged hepatectomy （RALPPS）.Investigators hypothesized that the RALPPS might result in lower morbidity and mortality rate than ALPPS in the treatment of hepatocellular carcinoma . This Prospective Randomized Controlled Trial is on the Safety and Efficacy of radio-frequency assisted liver partition with portal vein ligation for staged hepatectomy for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* An insufficient future liver remnant(FLR<30% in normal hepatic function or FLR<40% with hepatic cirrhosis or after chemotherapy）
* Liver function of Child-Pugh Class A or B.
* Liver Reserve Function：ICG-R15≤10％
* No evidence of coagulopathy: platelet count > 50 × 109/L and a prolonged prothrombin time of < 5 seconds.

Exclusion Criteria:

* Patients met the inclusion criteria but declined to participate.
* Patients with severe portal hypertension, a history of esophageal variceal hemorrhage, severe hypersplenism syndrome, or refractory ascites.
* Main portal vein、inferior vena cava、common hepatic duct and hepatic vein have tumor thrombus.
* Extrahepatic or lymph node metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
morbidity during perioperation | 2 years
  complications include bile leakage, abdominal infection, hemorrhage, PHLF e.t.
mortality during perioperation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China